CLINICAL TRIAL: NCT02580136
Title: Esthesioneuroblastoma: Outcomes After Treatment
Acronym: ENB
Status: Withdrawn | Type: Observational
Why Stopped: Lack of accrual
Sponsor: Ricardo L. Carrau, MD (Other)
Responsible Party: Sponsor-Investigator, Ricardo L. Carrau, MD, Ricardo L. Carrau, MD, Ohio State University
Organization: Ohio State University (Other)
Other Study IDs: 2015C0066
Record Dates: First submitted 2015-09-13; First posted 2015-10-20 (Estimated); Last update posted 2021-02-11 (Actual); Status verified 2021-02

CONDITIONS: Esthesioneuroblastoma, Olfactory
Keywords: Esthesioneuroblastoma; Tumor; Skull Base Surgery; Sinonasal Cancer
MeSH Terms: conditions — Esthesioneuroblastoma, Olfactory; Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 120 Months
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this study is to collect and organize data into a repository to gather relevant information for future research from patients diagnosed with a rare malignant sinonasal cancer called esthesioneuroblastoma (ENB) and are scheduled to undergo endonasal skull base surgery. Data being collected includes surgical data, demographics, disease presentation, MRI, CT, PET imaging, and post-operative assessments including pathology tests. After surgery, the investigators will collect chemotherapy and radiation data. Participants will also complete quality of life questionnaires at their follow-up visits.

ELIGIBILITY:
Inclusion Criteria:

* Between the age of 10-80 years
* Diagnosed with esthesioneuroblastoma

Exclusion Criteria:

* Refusal to participate

Ages: 10 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients diagnosed with esthesioneuroblastoma (ENB)
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2015-09; Primary Completion 2021-02-08 (Actual); Study Completion 2021-02-08 (Actual)

PRIMARY OUTCOMES:
Quality of Life | up to 120 months after treatment
  Anterior Skull Base (ASB); Skull Base Inventory (SBI); Multidimensional Disease Specific Inventory MDS; ASB-Nasal 12; Sino-Nasal Outcome Test (SNOT-20)
Progression-free survival and overall survival | Up to 120 months
  Kaplan-Meier survival curves

SECONDARY OUTCOMES:
Number of participants with intraoperative complications | up to 120 months
Number of participants with postoperative complications | up to 120 months
Length of Hospital Stay | up to 120 months
Time spent in operating room | up to 120 months
MRI imaging evidence of resection | up to 120 months
Surgical Technique | up to 120 months

CONTACTS AND LOCATIONS:
Overall Officials: Ricardo Carrau, MD, Principal Investigator — Ohio State University
Locations (1):
- The Ohio State University, Columbus, Ohio, United States